CLINICAL TRIAL: NCT06957210
Title: Post-Traumatic Growth Following Eye Movement Desensitization and Reprocessing Therapy Versus SSRIs in Patients With Post-Traumatic Stress Disorder: A Randomized Controlled Trial
Brief Title: Post-Traumatic Growth Following Eye Movement Desensitization and Reprocessing Therapy Versus SSRIs in Patients With Post-Traumatic Stress Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asad Ullah Jan (Other Government)
Collaborators: CMH Nowshera (Unknown)
Responsible Party: Sponsor-Investigator, Asad Ullah Jan, Head Department of Psychiatry, Combined Military Hospital Nowshera
Organization: Combined Military Hospital Nowshera (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMHNSR-REF-15
Record Dates: First submitted 2025-04-26; First posted 2025-05-04 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: PTSD - Post Traumatic Stress Disorder
Keywords: PTSD; Post-traumatic Stress Disorder; Post-traumatic Growth; EMDR; Eye Movement Desensitization and Reprocessing
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic | interventions — Eye Movement Desensitization Reprocessing; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMDR (Experimental): EMDR therapy
  Interventions: Behavioral: EMDR
- SSRIs (Active Comparator): Acting as control group
  Interventions: Drug: SSRIs

INTERVENTIONS:
Behavioral: EMDR — Participants will receive structured EMDR therapy sessions conducted by trained therapists following standard EMDR protocols. Sessions will occur weekly over a 6 week period.
  Arms: EMDR
Drug: SSRIs — Participants will receive pharmacotherapy with an SSRI prescribed according to standard clinical guidelines for PTSD, monitored by a psychiatrist over a 6-week period.
  Arms: SSRIs

SUMMARY:
This randomized controlled trial investigates the comparative effectiveness of Eye Movement Desensitization and Reprocessing (EMDR) therapy and selective serotonin reuptake inhibitors (SSRIs) in fostering post-traumatic growth among patients diagnosed with post-traumatic stress disorder (PTSD). Participants will be randomized to receive either EMDR therapy or standard SSRI pharmacotherapy. The primary objective is to evaluate the extent of psychological growth and recovery achieved through each intervention, aiming to guide future therapeutic strategies for PTSD.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Post-Traumatic Stress Disorder (PTSD) based on DSM-5 criteria

Willingness to participate and provide informed consent

Ability to comply with study procedures

Exclusion Criteria:

Current diagnosis of psychotic disorder, bipolar disorder, or severe major depressive episode with psychotic features

Active substance use disorder within the past 6 months

Severe cognitive impairment or inability to complete study assessments

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-Traumatic Growth (PTG) measured by Post-Traumatic Growth Inventory (PTGI) | 6 weeks
  Change in PTGI total score from baseline to 6 weeks.

SECONDARY OUTCOMES:
PTSD symptom severity measured by PTSD Checklist | 6 weeks
  Change in PTSD Checklist total score from baseline to 6 weeks.

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Combined Military Hospital, Nowshera, KPK
  - Department of Psychiatry, Combined Military Hospital Nowshera, Nowshera, KPK

IPD SHARING:
Plan to Share IPD: No
Privacy concerns and confidentiality protections for participants limit the feasibility of public data sharing.